CLINICAL TRIAL: NCT01994876
Title: Investigation of Newly Developed 1-piece Convex Baseplates in Subjects With Ileostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CP229
Record Dates: First submitted 2013-10-01; First posted 2013-11-26 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-02

CONDITIONS: Ileostomy - Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- First Coloplast Test 1 (Experimental): The subjects first test their own product to collect a baseline measurement
  The subjects are randomised to first test Coloplast Test 1 and thereafter Coloplast Test 2
  Interventions: Device: Coloplast Test 1; Device: Coloplast Test 2
- First Coloplast Test 2 (Experimental): The subjects first test their own product to collect baseline measurements
  The subjects are randomised to first test Coloplast Test 2 and thereafter Coloplast Test 1
  Interventions: Device: Coloplast Test 1; Device: Coloplast Test 2

INTERVENTIONS:
Device: Coloplast Test 1 — Coloplast Test 1 is a newly developed 1-piece convex ostomy appliance
Device: Coloplast Test 2 — Coloplast Test 2 is a newly developed 1-piece convex ostomy appliance

SUMMARY:
To investigate the performance and safety of two newly developed convex 1-piece ostomy appliances

ELIGIBILITY:
Inclusion Criteria:

Subjects must comply with the following criteria in order to participate in the investigation:

1. Are at least 18 years of age and have full legal capacity
2. Have had an ileostomy for at least 3 months
3. Have used a convex ostomy appliance for the last month
4. Have given written informed consent
5. Have an ileostomy with a diameter of 33 mm or less
6. Have experience leakage (seeping) under the baseplate at least two times over the last two weeks

Exclusion Criteria:

Subjects complying with the following criteria must be excluded from participation in the clinical investigation:

1. Have a loop ostomy (also called double-barrel or ostomy with two outlets)
2. Are pregnant or breastfeeding
3. Currently receiving, or have received within the last 2 months, chemotherapy or radiation therapy.
4. Currently receiving or have received, within the last month, systemic or local steroid treatment (adreno-cortical hormone) in the peristomal area
5. Currently suffering from peristomal skin problems (i.e. bleeding or broken skin (weeping skin))
6. Are currently participating in another clinical investigation or has previously participated in this investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kalid S Abd-Elaziz, MD, Principal Investigator — QPS Holdings LLC
Locations (1):
- QPS, Groningen, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subject were recruited through the Coloplast database in The Netherlands
Groups:
- First Coloplast Test 1, Then Coloplast Test 2: The subjects first test their own product to collect a baseline measurement
  The subjects are randomised to first test Coloplast Test 1 and thereafter Coloplast Test 2
  Coloplast Test 1: Coloplast Test 1 is a newly developed 1-piece convex ostomy appliance
  Coloplast Test 2: Coloplast Test 2 is a newly developed 1-piece convex ostomy appliance
- First Coloplast Test 2, Then Coloplast Test 1: The subjects first test their own product to collect baseline measurements
  The subjects are randomised to first test Coloplast Test 2 and thereafter Coloplast Test 1
  Coloplast Test 1: Coloplast Test 1 is a newly developed 1-piece convex ostomy appliance
  Coloplast Test 2: Coloplast Test 2 is a newly developed 1-piece convex ostomy appliance
Period: Baseline - Own Product
Arm/Group | First Coloplast Test 1, Then Coloplast Test 2 | First Coloplast Test 2, Then Coloplast Test 1
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Test Period 1
Arm/Group | First Coloplast Test 1, Then Coloplast Test 2 | First Coloplast Test 2, Then Coloplast Test 1
Started | 9 | 9
Completed | 9 | 7
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Test Period 2
Arm/Group | First Coloplast Test 1, Then Coloplast Test 2 | First Coloplast Test 2, Then Coloplast Test 1
Started | 9 | 7
Completed | 8 | 6
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: All the subjects in one group
Arm/Group | Overall Study
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Degree of Leakage
Description: The degree of leakage was measured with a 32-point scale developed by Coloplast A/S, where 0 point represents the best possible outcome (no leakage) and 32 represents the worst possible outcome (full leakage under baseplate)
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: baseplates
Groups:
- Coloplast Test 1: Results from subjects testing Coloplast Test 1
- Coloplast Test 2: Results from subjects testing Coloplast Test 2
- Basline - Own Product: Data from subject testing own product. Measures baseline leakage
Arm/Group | Coloplast Test 1 | Coloplast Test 2 | Basline - Own Product
Number analyzed (Participants) | 16 | 18 | 18
Number analyzed (baseplates) | 229 | 208 | 267
units on a scale | 1.9 (4.2) | 2.5 (4.3) | 3.1 (5.7)

ADVERSE EVENTS:
Time Frame: September - November 2012
Arm/Group | Coloplast Test 1 | Coloplast Test 2 | Basline - Own Product
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 3/16 | 1/18 | 0/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coloplast Test 1 (N=16) | Coloplast Test 2 (N=18) | Basline - Own Product (N=18)
Redness skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Peristomal skin irritaion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes